CLINICAL TRIAL: NCT02946736
Title: Evaluation of a Work-Family and Sleep Leadership Intervention in the Oregon National Guard: A Behavioral Health Leadership Approach
Brief Title: Oregon Military Employee Sleep and Health Study
Acronym: MESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland State University (Other); Colorado State University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Hammer, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: W81XWH-16-1-0720
Record Dates: First submitted 2016-10-19; First posted 2016-10-27 (Estimated); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Well-Being; Sleep; Health Behavior
Keywords: Sleep; Physical Health; Psychological Health; Well-Being; Employee; Actigraphy
MeSH Terms: conditions — Health Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervisor Intervention (Experimental): Supervisors in the intervention group will go through the FSSB/sleep leadership training and receive actigraphy feedback.
  Interventions: Behavioral: FSSB/Sleep Leadership Training; Behavioral: Actigraphy Feedback
- Employee Intervention (Experimental): Employees in the intervention group will receive actigraphy feedback.
  Interventions: Behavioral: Actigraphy Feedback
- Waitlist Control (No Intervention): Supervisor training and actigraphy feedback provided AFTER final 9 month data collection.

INTERVENTIONS:
Behavioral: FSSB/Sleep Leadership Training — Supervisors will receive a training addressing family-supportive supervisor behaviors and sleep leadership.
  Arms: Supervisor Intervention
Behavioral: Actigraphy Feedback — Supervisors and employees will receive personalized feedback on their sleep and activity measurements.
  Arms: Employee Intervention; Supervisor Intervention

SUMMARY:
This study is a randomized controlled trial that assesses the effects of (1) the Family-Supportive Supervisor Behavior (FSSB) and Sleep Leadership training and (2) sleep/cognitive effectiveness feedback intervention on health and well-being among full-time employees in the Oregon National Guard, their supervisors, and their families. The interventions involving both health protection and health promotion are expected to contribute to improvements in employees' and their supervisors' sleep, risk behaviors, mental and physical health, and injury, as well as employees' and their spouse/partners' family experiences, health and well-being, and workplace outcomes.

DETAILED DESCRIPTION:
The overall goal of the Military Employee Sleep and Health (MESH) study is to improve safety, health and well-being of service members in the Oregon National Guard and their families. The MESH Study seeks to do this by training supervisors to support Oregon National Guard service members by focusing on a reduction in work-life stress while increasing sleep health.

The Oregon MESH Study proposes that leadership can influence a fundamental change in the recognition of sleep health and service members' overall well-being and the well-being of their family members. With the support of the Oregon National Guard, the MESH Study will provide family-support and sleep leadership training for supervisors while raising awareness of sleep through daily non-invasive sleep measurements.

The investigators of the Oregon MESH Study expect positive results for study participants, including reduced stress and increased social support. Longer term, these effects are expected to create a more supportive work environment, which has positive effects on safety, health, well-being, family, and organizational outcomes. The investigators also expect that providing service members with individual sleep feedback will reduce sleep problems and improve sleep awareness.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees in the Oregon National Guard, including Military Technicians and Active Guard Reserves.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hammer, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hobfoll, S. E., Vinokur, A. D., Pierce, P. F., & Lewandowski-Romps, L. (2012). The combined stress of family life, work, and war in Air Force men and women: A test of conservation of resources theory. International Journal of Stress Management, 19(3), 217-237.
- See also: Sleep Disturbance Scale — http://www.healthmeasures.net/administrator/components/com_instruments/uploads/PROMIS%20SF%20v1.0%20-%20Sleep%20Disturbance%208b%205-3-20126.pdf
- See also: Sleep-Related Impairment Scale — http://www.healthmeasures.net/administrator/components/com_instruments/uploads/PROMIS%20SF%20v1.0%20-%20Sleep%20Related%20Impairment%20%208a%205-9-2016.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n=215 were identified as supervisors in the intervention condition and were excluded (i.e., focus is on service members only for analysis)
Groups:
- Intervention Combined: Service Member/Employees: Includes all service members/employees who are in the intervention condition, which includes both treatments: 1) Their supervisor is in the condition for the Sleep Leadership/Family Supportive training and 2) the service member is in the sleep actigraphy feedback condition.
- Waitlist Control: Service members do not receive actigraphy feedback nor do their supervisors receive the sleep leadership/Family Supportive training until AFTER final data collection at 9 months
Period: Employees: 4 Month Completion
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Started | 358 | 346
Completed | 295 | 289
Not Completed | 63 | 57
Period: Employees: 9 Month Completion
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Started | 295 | 289
Completed | 275 | 274
Not Completed | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Intervention Combined: Service Member/Employees: Includes all service members/employees who are in the intervention condition, which includes both treatments: 1) Their supervisor is in the condition for the Sleep Leadership/FSSB training and 2) the service member is in the sleep actigraphy feedback condition.
- Waitlist Control: Service members do not receive actigraphy feedback NOR do their supervisors receive the sleep leadership/FSSB training until AFTER final data collection at 9 months
- Total: Total of all reporting groups
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control | Total
Number analyzed (Participants) | 358 | 346 | 704
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.94 (8.98) | 36.49 (9.18) | 36.21 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 357 | 346 | 703
    Female | 90 | 87 | 177
    Male | 267 | 259 | 526
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    Dichotomized Race/Ethnicity: number analyzed (Participants) | 356 | 344 | 700
    Dichotomized Race/Ethnicity: White | 289 | 276 | 565
    Dichotomized Race/Ethnicity: Non-White/Multiple | 67 | 68 | 135
Region of Enrollment [Number; unit: participants]
  United States | 358 | 346 | 704
Self-Reported Sleep Duration [Mean (Standard Deviation); unit: Hours] — Total number of hours calculated from reported bed time and wake time. Source: Buysse et al., 1989
  Hours | 7.29 (1.09) | 7.28 (1.06) | 7.28 (1.08)
Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Disturbance Insomnia Subsca [Mean (Standard Deviation); unit: units on a scale] — Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much).
  T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured (worse).
  units on a scale | 52.47 (8.52) | 52.79 (7.86) | 52.63 (8.20)
Patient Reported Outcomes Measurement Information System (PROMIS): Dissatisfaction With Sleep Subsca [Mean (Standard Deviation); unit: units on a scale] — Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much.
  T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured (worse).
  units on a scale | 53.88 (7.68) | 54.08 (7.33) | 53.98 (7.51)
Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Related Impairment Subscale [Mean (Standard Deviation); unit: units on a scale] — 8 item scale. Likert-type responses: 1 = Not at all to 5 = Very much). T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more sleep impairment (worse).
  units on a scale | 53.07 (8.85) | 53.35 (8.40) | 53.21 (8.63)
Actigraphic Sleep Duration: Total Sleep Time (TST) [Mean (Standard Deviation); unit: Hours] — Actigraphic measurements obtained using Actiwatch2 worn for 3 weeks Average sleep duration in hours Great duration generally better, with target range of 7-9 hours each sleep period.
  Hours | 6.61 (.77) | 6.59 (.80) | 6.60 (.79)
Actigraphic Sleep Efficiency: Wake After Sleep Onset (WASO) [Mean (Standard Deviation); unit: Minutes] — Actigraphic measurements obtained using Actiwatch2 worn for 3 weeks Average number of minutes spent awake during the sleep period. More minutes indicates worse outcome.
  Minutes | 41.06 (12.03) | 41.31 (12.81) | 41.19 (12.42)
Overall Job Satisfaction Scale [Mean (Standard Deviation); unit: units on a scale] — Service member satisfaction with current job; Likert-type scale 1 = Strongly disagree to 5 = Strongly agree, mean created from the 3 items.
  Scores could range from 0-5 with higher levels indicating greater satisfaction. Source: Cammann et al., 1983
  units on a scale | 3.98 (.85) | 3.90 (.85) | 3.94 (.85)
Turnover Intentions [Mean (Standard Deviation); unit: units on a scale] — Service member intention to quit current job; Two items with responses on Likert-type scale 1 = Strongly disagree to 5 = Strongly agree.
  Overall score created with a mean of the two items, with higher levels indicating greater intention to leave one's job.
  Source: Boroff & Lewin, 1997
  units on a scale | 2.04 (1.15) | 2.23 (1.23) | 2.13 (1.19)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — Service member self-reported stress; Likert-type scale 0 = Never to 4 = Very often, combined to a mean score, with a possible range from 0 to 4.
  Higher scores indicate greater stress (worse). Source: Cohen & Williamson, 1988
  units on a scale | 1.37 (.70) | 1.37 (.67) | 1.37 (.68)
Walter Reed Functional Impairment: Occupational Subscale (OFI) [Mean (Standard Deviation); unit: units on a scale] — Service member difficulty with completing work tasks and quality; 6 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
  units on a scale | 1.83 (.82) | 1.79 (.73) | 1.81 (.78)
Walter Reed Functional Impairment: Social Functional Impairment (SFI) [Mean (Standard Deviation); unit: units on a scale] — Service member difficulty functioning in social situations; 4 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
  units on a scale | 1.68 (.66) | 1.69 (.67) | 1.68 (.66)
Walter Reed Functional Impairment: Personal Functional Impairment (PFI) [Mean (Standard Deviation); unit: units on a scale] — Service member difficulty with getting personal life skills completed; 2 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
  units on a scale | 1.60 (.75) | 1.63 (.76) | 1.61 (.76)

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Sleep Duration
Description: Total number of hours calculated from reported bed time and wake time. Minimum 0 hours, Maximum 24 hours. Longer duration indicates longer sleep duration. Ideal range is 7-9 hours of sleep per night.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 270 | 271
Hours | 7.43 (1.10) | 7.34 (1.13)

2. Primary Outcome: Self-Reported Sleep Duration
Description: as for outcome 1
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 251 | 260
Hours | 7.50 (1.15) | 7.39 (1.21)

3. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Disturbance Insomnia Subscale
Description: Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much).
  T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. This is considered the most accurate option.
  T-Scores estimates were developed using a population of 2,252 participants, 259 of which had clinical sleep disorders, and was intended to be representative of the US population. This is the reference population that the T-score means and SDs were calibrated and centered with.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured (worse).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 269 | 272
t score on a scale | 50.90 (8.65) | 51.78 (8.01)

4. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Disturbance Insomnia Subscale
Description: Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much). T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. This is considered the most accurate option.
  T-Scores estimates were developed using a population of 2,252 participants, 259 of which had clinical sleep disorders, and was intended to be representative of the US population. This is the reference population that the T-score means and SDs were calibrated and centered with.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 251 | 260
t score on a scale | 51.63 (8.48) | 52.00 (8.21)

5. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Dissatisfaction With Sleep Subscale
Description: Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much.
  T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. This is considered the most accurate option.
  T-Scores estimates were developed using a population of 2,252 participants, 259 of which had clinical sleep disorders, and was intended to be representative of the US population. This is the reference population that the T-score means and SDs were calibrated and centered with.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured (worse).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 269 | 272
t score on a scale | 52.28 (8.06) | 53.27 (7.98)

6. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Dissatisfaction With Sleep Subscale
Description: Four item subscale of the larger 8 item Sleep Disturbance scale. Likert-type responses: 1 = Not at all to 5 = Very much).
  T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. This is considered the most accurate option.
  T-Scores estimates for Dissatisfaction with Sleep were developed using a population of 2,252 participants, 259 of which had clinical sleep disorders, and was intended to be representative of the US population. This is the reference population that the T-score means and SDs were calibrated and centered with.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more of the concept being measured (worse).
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 251 | 259
t score on a scale | 52.26 (7.79) | 53.32 (7.68)

7. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Related Impairment Subscale (SRI)
Description: 8 item scale. Likert-type responses: 1 = Not at all to 5 = Very much). T-Scores were created using HealthMeasures Scoring service, where data are uploaded into the HealthMeasures scoring service website, which generates T-Scores. This is considered the most accurate option.
  T-Scores estimates for SRI were developed using a population of 2,252 participants, 259 of which had clinical sleep disorders, and was intended to be representative of the US population. This is the reference population that the T-score means and SDs were calibrated and centered with.
  The T-Scores that HealthMeasures generates are not precisely at a mean of 50 and standard deviation of 10 because they are based on the unique MESH samples. A higher PROMIS T-score represents more sleep impairment (worse).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 270 | 272
t score on a scale | 51.10 (9.58) | 52.33 (8.66)

8. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS): Sleep Related Impairment Subscale (SRI)
Description: as for outcome 7
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: t score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 251 | 260
t score on a scale | 50.91 (9.12) | 51.91 (8.33)

9. Primary Outcome: Actigraphic Sleep Duration: Total Sleep Time (TST)
Description: Actigraphic measurements obtained using Actiwatch2 worn for 3 weeks Average sleep duration in hours Great duration generally better, with target range of 7-9 hours each sleep period.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 227 | 256
Hours | 6.65 (.79) | 6.54 (.96)

10. Primary Outcome: Actigraphic Sleep Efficiency: Wake After Sleep Onset (WASO)
Description: Actigraphic measurements obtained using Actiwatch2 worn for 3 weeks Average number of minutes spent awake during the sleep period. More minutes indicates worse outcome.
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 227 | 253
Minutes | 42.76 (13.90) | 42.71 (13.73)

11. Primary Outcome: Overall Job Satisfaction Scale
Description: Service member satisfaction with current job; Likert-type scale 1 = Strongly disagree to 5 = Strongly agree, mean created from the 3 items.
  Scores could range from 0-5 with higher levels indicating greater satisfaction. Source: Cammann et al., 1983
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 261 | 262
score on a scale | 3.86 (.82) | 3.80 (.94)

12. Primary Outcome: Turnover Intentions
Description: Service member intention to quit current job; Two items with responses on Likert-type scale 1 = Strongly disagree to 5 = Strongly agree.
  Overall score created with a mean of the two items, with higher levels indicating greater intention to leave one's job.
  Source: Boroff & Lewin, 1997
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 259 | 263
score on a scale | 2.25 (1.00) | 2.32 (1.27)

13. Primary Outcome: Perceived Stress Scale
Description: Service member self-reported stress; Likert-type scale 0 = Never to 4 = Very often, combined to a mean score, with a possible range from 0 to 4.
  Higher scores indicate greater stress (worse). Source: Cohen & Williamson, 1988
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 253 | 260
score on a scale | 1.35 (.71) | 1.38 (.67)

14. Primary Outcome: Walter Reed Functional Impairment: Occupational Subscale (OFI)
Description: Service member difficulty with completing work tasks and quality; 6 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 252 | 259
score on a scale | 1.79 (.77) | 1.73 (.76)

15. Primary Outcome: Walter Reed Functional Impairment Scale: Personal Functioning Subscale (PFI)
Description: Service member difficulty with getting personal life skills completed; 2 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 253 | 260
score on a scale | 1.66 (.67) | 1.68 (.69)

16. Primary Outcome: Walter Reed Functional Impairment Scale: Social Functional Impairment Subscale (SFI)
Description: Service member difficulty functioning in social situations; 4 items with Likert-type responses: 1 = No difficulty at all to 5 = Extreme difficulty, mean score created from all items, with possible score range from 1 to 5.
  Higher levels indicating greater impairment (worse). Source: Subscale of Overall Functional Impairment by Herrell et al., 2014
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 252 | 256
score on a scale | 1.55 (.70) | 1.54 (.68)

17. Secondary Outcome: Family Supportive Supervisor Behaviors (FSSB)
Description: Perceived supervisor support for work-family integration as reported by service member, 4 items, with responses on Likert-type scale 1=Strongly disagree to 5= Strongly agree, overall score created by mean score, with possible scores ranging from 1 to 5..
  Higher scores indicating higher levels of support (better) Source: Hammer et al., 2013
Time Frame: 4-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 286 | 283
score on a scale | 4.12 (.91) | 3.98 (.94)

18. Secondary Outcome: Sleep Leadership
Description: Perceived supervisor support for sleep health as reported by service member, 8 items, with responses on Likert-type scale 1=Never to 5= Always, overall score created by mean score, with possible scores ranging from 1 to 5..
  Higher scores indicating higher levels of support (better) Source: Modified version of Gunia et al., 2015
Time Frame: 4-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
Number analyzed (Participants) | 283 | 284
score on a scale | 2.54 (1.05) | 2.32 (.95)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Minimal risk protocol
Arm/Group | Intervention Combined: Service Member/Employees | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/358 | 0/346
Serious Adverse Events (participants affected / at risk) | 0/358 | 0/346
Other Adverse Events (participants affected / at risk) | 0/358 | 0/346

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02946736/Prot_SAP_000.pdf